CLINICAL TRIAL: NCT07257445
Title: Comparative Study Between Different Surgical Modalities in Management of Severe Grades of Gynecomastia.
Brief Title: Modularities of Management of Severe Grades of Gynecomastia.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Mohamed Hassan, Assistant Lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Severe grades of Gynecomastia
Record Dates: First submitted 2025-11-16; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Gynecomastia
Keywords: Severe Gynecomastia; Management of gynecomastia
MeSH Terms: conditions — Gynecomastia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A: circumerolar skin excision (Experimental): Group A:
  1. We normally outline a 30-mm-diameter nipple-areola complex around the existing nipple.
  2. A second complete circumareolar circle representing the epidermal ring to be deepithelialized, the diameter is adapted in all direction (upper, lower, lateral and medial pole)to achieve the presence of the new NAC in the 4th intercostal space at mid clavicular line .
  Surgical procedure:
  * Under general anesthesia, patient is in supine position on the operation room table.
  * After marking the incisions and new nipple position, the areola was slightly stretched and marked with a 3 cm cookie cutter.
  * The complete circumareolar ring is deepithelialized.
  * An incision is then made from 3 o'clock to 9 o'clock along the inferior border of the deepithelialized ring.
  * Subcutaneous glandular excision is completed through that incision.
  * a closed suction drain is then placed.
  * A 3-0 polypropylene intradermal circumareolar purse string suture is used for skin closure.
  * Fe
  Interventions: Procedure: Group A: circumerolar skin excision
- Group B: elliptical skin excision with pedicled flap +/- lateral roll excision. (Experimental): Group B:
  1. The sternal notch with the mid sternal line, the inframammary crease line and the mid breast line.
  2. The new nipple position is located on the 4th intercostal space MCL.
  3. The mid breast line is marked from the clavicle to the nipple and then continued from the inframammary crease down the lower thoracic wall.
  4. the new inframammary fold is in the 6th intercostal space about 2-3 cm beneath the ideal NAC position.
  5. Within this marking the inferior pedicle is designed starting from the NAC apex down to the actual inferior mammary fold. The base of the inferior pedicle should not measure less than 6cm.
     The excised part marked as an elliptical excision between the actual and ideal inframammary fold with extension to the lateral roll if present.
  6. The symmetry of the markings, especially the new NAC positions, are checked in front of a mirror.
  Interventions: Procedure: Group B: elliptical skin excision with pedicled flap +_ lateral roll excision.
- Group C: elliptical skin excision with free nipple areola complex +/_ lateral roll excision. (Experimental): Group C:
  1. The sternal notch with the mid sternal line, the inframammary crease line and the mid breast line.
  2. The new nipple position is located on the 4th intercostal space MCL.
  3. The mid breast line is marked from the clavicle to the nipple and then continued from the inframammary crease down the lower thoracic wall.
  4. the ideal inframammary fold is in the 6th intercostal space about 2-3 cm beneath the ideal NAC position.
  5. The excised part marked as an elliptical excision between the actual and ideal inframammary fold with extension to the lateral roll if present.
  6. The symmetry of the markings, especially the new NAC positions, are checked in front of a mirror.
     * After marking, the nipple areola complex will be taken as a full thickness graft
     * The excisable part will be excised and restitched by 2\0 vicryl subcutaneously and 3\0 vicryl subcuticular sutures.
     * the recipient site of the NAC is deepithelized and the graft will be insit with tie-over for 1 week.
  Interventions: Procedure: Group C: elliptical skin excision with free nipple areola complex +_ lateral roll excision.

INTERVENTIONS:
Procedure: Group A: circumerolar skin excision — Surgical procedure:
  * Under general anesthesia, patient is in supine position on the operation room table.
  * After marking the incisions and new nipple position, the areola was slightly stretched and marked with a 3 cm cookie cutter.
  GROUP A:
  * The complete circumareolar ring is deepithelialized.
  * An incision is then made from 3 o'clock to 9 o'clock along the inferior border of the deepithelialized ring.
  * Subcutaneous glandular excision is completed through that incision.
  * a closed suction drain is then placed.
  * A 3-0 polypropylene intradermal circumareolar purse string suture is used for skin closure.
  * Few interrupted 5-0 absorbable sutures are also used to adjust skin edges at the purse string closure.
  * An elastic compressive garment is applied intraoperatively and is worn for 6 weeks.
  Arms: Group A: circumerolar skin excision
Procedure: Group B: elliptical skin excision with pedicled flap +_ lateral roll excision. — GROUP B:
  * Following marking, epithelialization of the inferior pedicle flap is performed. The excisable tissue is then resected, and the pedicle is carefully dissected down to the pectoral fascia.
  * Flap thinning is carried out cautiously, preserving the dermis and a thin layer of subcutaneous tissue to maintain vascularity. A subcutaneous tunnel is subsequently created towards the new NAC site by excising the intervening adipose tissue, allowing for proper transposition of the pedicle.
  * After preparation of the tunnel, the inferior pedicle is transposed into the new nipple-areola complex (NAC) site. The pedicle is secured in place with interrupted non-absorbable sutures to prevent displacement and to maintain adequate projection.
  * The NAC is then inset into the newly created pocket, ensuring symmetry and central positioning. Excess skin and redundant tissue are trimmed as required to optimize chest contour.
  * The wound is closed in layers using deep absorbable sutures for support
  Arms: Group B: elliptical skin excision with pedicled flap +/- lateral roll excision.
Procedure: Group C: elliptical skin excision with free nipple areola complex +_ lateral roll excision. — GROUP C:
  * After marking, the nipple areola complex will be taken as a full thickness graft
  * The excisable part will be excised and restitched by 2\0 vicryl subcutaneously and 3\0 vicryl subcuticular sutures.
  * the recipient site of the NAC is deepithelized and the graft will be insit with tie-over for 1 week and the drain inserted for 4-7 days
  Arms: Group C: elliptical skin excision with free nipple areola complex +/_ lateral roll excision.

SUMMARY:
Gynecomastia is defined as a benign enlargement of the mammary glands, commonly diffused among men. The prevalence of gynecomastia ranges from 38 to 64 percent in the male population.

Gynecomastia can affect normal self-esteem and sexual identity and often patients feel ashamed of their bodies during normal social activities.

The surgical management of the high-grade gynecomastia Simon's grade III or Rohrich's grade IV has remained problematic because both liposuction and conventional subcutaneous mastectomy without skin excision have frequently resulted in significant residual skin redundancy, requiring a second operation for skin resection.

Two Classification Systems of Gynecomastia

Rohrich's Classification I, Minimal breast hypertrophy without ptosis; hypertrophy is either primarily glandular or fibrous II, Moderate breast hypertrophy without ptosis; hypertrophy is either primarily glandular or fibrous III, Severe breast hypertrophy with grade I ptosis glandular or fibrous IV, Severe breast hypertrophy with grade II or III ptosis glandular or fibrous Simon's Classification I, Minor breast enlargement without skin redundancy. IIa, Moderate breast enlargement without skin redundancy IIb, Moderate breast enlargement with minor skin redundancy III, Gross breast enlargement with skin redundancy that simulates a pendulous female breast Smoot stated that this approach for high-grade gynecomastia has several disadvantages. There are difficulties in obtaining precertification from third-party payers for a second operation for skin resection. In addition, the adolescent patient is often very anxious during the ensuring 1 year after the original mastectomy when skin excess is quite apparent and awaiting spontaneous shrinkage.

Currently, there are 4 main different approaches for the management of high-grade gynecomastia:

First is simple mastectomy, which is done with free nipple graft accepting the long transverse scar and the grafted appearance of the nipple areola complex. Second is a modification of breast reduction is done with nipple transposition on a single dermal pedicle or vertical bipedicle. A visible chest scar is also present, but the blood supply of the nipple-areola complex is preserved.

Third is ultrasound assisted liposuction is performed first and after several months, accept that several patients will require a second operation to excise the significant residual skin redundancy. Fourth is a single-stage procedure is done in which sub cutaneous mastectomy and circumareolar skin excision are performed. The purse string skin closure limits the scar to the circumareolar area.

Open excision techniques base their principle on a direct view and management of the gland, through several types of surgical accesses according to the surgeon's preference and entity of the defect. The main advantage of open excision is the direct control of the hemostasis and redundant skin control, with the main disadvantage of permanent scars, whose quality cannot be predicted.

Only Gusenoff et al have proposed a classification with corresponding operative treatment options, whose grades taken into account the laxity of the breast skin and the upper abdomen, the location of the inframammary fold IMF, and the lateral fat role.

Minimal excess skin and fat, minimal alteration of NAC, normal IMF, No lateral skin roll: a Minimal excess skin and fat, minimal alteration of NAC, normal IMF, lateral skin roll: b NAC and IMF below, the ideal IMF, lateral chest roll, minimal upper abdominal laxity: c NAC and IMF below the ideal IMF, lateral chest roll, significant upper abdominal laxity: d

DETAILED DESCRIPTION:
Cases will be divided into 3 groups according to skin incision:

Group A: circumerolar skin excision Group B: elliptical skin excision with pedicled flap +_ lateral roll excision. Group C: elliptical skin excision with free nipple areola complex +_ lateral roll excision.

Markings

-The preoperative drawings proceed with the patient in standing position.

Group A:

1. We normally outline a 30-mm-diameter nipple-areola complex around the existing nipple.
2. A second complete circumareolar circle representing the epidermal ring to be deepithelialized, the diameter is adapted in all direction (upper, lower, lateral and medial pole)to achieve the presence of the new NAC in the 4th intercostal space at mid clavicular line .

Group B:

1. The sternal notch with the mid sternal line, the inframammary crease line and the mid breast line.
2. The new nipple position is located on the 4th intercostal space MCL.
3. The mid breast line is marked from the clavicle to the nipple and then continued from the inframammary crease down the lower thoracic wall.
4. the new inframammary fold is in the 6th intercostal space about 2-3 cm beneath the ideal NAC position.
5. Within this marking the inferior pedicle is designed starting from the NAC apex down to the actual inferior mammary fold. The base of the inferior pedicle should not measure less than 6cm.

   The excised part marked as an elliptical excision between the actual and ideal inframammary fold with extension to the lateral roll if present.
6. The symmetry of the markings, especially the new NAC positions, are checked in front of a mirror.

Group C:

1. The sternal notch with the mid sternal line, the inframammary crease line and the mid breast line.
2. The new nipple position is located on the 4th intercostal space MCL.
3. The mid breast line is marked from the clavicle to the nipple and then continued from the inframammary crease down the lower thoracic wall.
4. the ideal inframammary fold is in the 6th intercostal space about 2-3 cm beneath the ideal NAC position.
5. The excised part marked as an elliptical excision between the actual and ideal inframammary fold with extension to the lateral roll if present.
6. The symmetry of the markings, especially the new NAC positions, are checked in front of a mirror.

Surgical procedure:

* Under general anesthesia, patient is in supine position on the operation room table.
* After marking the incisions and new nipple position, the areola was slightly stretched and marked with a 3 cm cookie cutter.

GROUP A:

* The complete circumareolar ring is deepithelialized.
* An incision is then made from 3 o'clock to 9 o'clock along the inferior border of the deepithelialized ring.
* Subcutaneous glandular excision is completed through that incision.
* a closed suction drain is then placed.
* A 3-0 polypropylene intradermal circumareolar purse string suture is used for skin closure.
* Few interrupted 5-0 absorbable sutures are also used to adjust skin edges at the purse string closure.
* An elastic compressive garment is applied intraoperatively and is worn for 6 weeks.

GROUP B:

* Following marking, epithelialization of the inferior pedicle flap is performed. The excisable tissue is then resected, and the pedicle is carefully dissected down to the pectoral fascia.
* Flap thinning is carried out cautiously, preserving the dermis and a thin layer of subcutaneous tissue to maintain vascularity. A subcutaneous tunnel is subsequently created towards the new NAC site by excising the intervening adipose tissue, allowing for proper transposition of the pedicle.
* After preparation of the tunnel, the inferior pedicle is transposed into the new nipple-areola complex (NAC) site. The pedicle is secured in place with interrupted non-absorbable sutures to prevent displacement and to maintain adequate projection.
* The NAC is then inset into the newly created pocket, ensuring symmetry and central positioning. Excess skin and redundant tissue are trimmed as required to optimize chest contour.
* The wound is closed in layers using deep absorbable sutures for support, followed by a fine subcuticular closure to achieve minimal scarring. Small suction drains may be inserted if necessary to reduce the risk of seroma or hematoma formation.
* Finally, a light compressive dressing is applied to maintain flap stability and reduce postoperative edema

GROUP C:

* After marking, the nipple areola complex will be taken as a full thickness graft
* The excisable part will be excised and restitched by 2-0 vicryl subcutaneously and 3\0 vicryl subcuticular sutures.
* the recipient site of the NAC is deepithelized and the graft will be insit with tie-over for 1 week and the drain inserted for 4-7 days

Postoperative Care

* A change of dressing is carried out after 48 hours.
* Skin stitches are usually absorbed within 3 weeks. Postoperatively.
* Patients are instructed to lie semi-sitting.

Post-operative data:

Breast measurements: the same measurements that were taken preoperatively. patient satisfaction level: which is measured using a questionnaire that have scored through points: completely dissatisfied, slightly dissatisfied, poorly satisfied, fairly satisfied, completely satisfied. aesthetic outcome, nipple sensation , nipple color ,scar satisfaction and muscular contour.

Nipple assessment : colour ,sensitivity and vascularity Scar assessment by VANCOUVER SCAR SCALE 6 months postoperative complication: early such as wound dehiscence, ischemia, hematoma and seroma. Late complications such as nipple pigmentation, nipple sensation, scar, aesthetic outcome.

Photographic Documentation: At the same positions taken preoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. Grade IIb, III gynecomastia according to Simon classification.
2. Age is between 18 years and 60 years old.
3. Stable weight in last 6 months Exclusion Criteria

1- Age is below 18 years and above 60 years. 2- Grade I and IIA gynecomastia according to Simon classification. 3- Psychological problems. 4- Non compliant patient. 5- Unstable weight in last 6 months

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — only male
Enrollment: 45 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
patients satisfaction score after operation | Six month.
  using satisfaction score
  1 completely dissatisfied, 2 slightly dissatisfied, 3 poorly satisfied, 4 fairly satisfied,5 completely satisfied.

SECONDARY OUTCOMES:
VANCOUVER SCAR SCALE | 6 month.
  (1) height and pliability; and (2) height, pliability, and vascularity. Of note, these combinations did not include the pigmentation sub-score, since pigmentation is scored on a nominal rather than an ordinal scale; i.e., hyperpigmentation (2 points) is not necessarily more severe than hypopigmentation (1 point).

IPD SHARING:
Plan to Share IPD: Undecided